CLINICAL TRIAL: NCT02175303
Title: A Pilot Study Using Placenta Derived Decidual Stromal Cells for Toxicity and Inflammation With Special Focus to the Allogeneic Hematopoietic Cell Transplantation Setting
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Olle Ringdén, Professor, Karolinska Institutet
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DSCINF001
Record Dates: First submitted 2014-06-24; First posted 2014-06-26 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-06

CONDITIONS: Acute Lung Injury; Decidual Stromal Cells; Stem Cell Transplantation; Inflammation
MeSH Terms: conditions — Acute Lung Injury; Inflammation

ARMS (1):
- Decidual stromal cell therapy for toxicity and inflammation (Experimental): Patients with toxicity, inflammation or hemorrhages will receive decidual stromal cells at approximately 1x10^6 cells/kg at one or more occasions at weekly intervals dependent on clinical response.
  Interventions: Biological: Decidual stromal cell therapy

INTERVENTIONS:
Biological: Decidual stromal cell therapy — Decidual stromal cells from placenta will be infused intravenously at approximately 1x10^6 cells/kg at one or more occasions at weekly intervals.

SUMMARY:
To evaluate safety and efficacy using decidual stromal cell therapy for toxicity and inflammation, with special focus on allogeneic hematopoietic cell transplantation patients. The hypothesis to be tested is that the cells are safe to infuse and that they have an anti-inflammatory and healing effect.

DETAILED DESCRIPTION:
Patients with toxicity, inflammation or hemorrhages will receive decidual stromal cells at approximately 1x10^6 cells/kg at one or more occasions at weekly intervals dependent on clinical response.

ELIGIBILITY:
Inclusion Criteria:

* Patients with toxicity, inflammation or hemorrhages.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2013-12; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Number of adverse events | Up to one year after inclusion

SECONDARY OUTCOMES:
Anti-inflammatory and reparatory effects regarding different lesions. | Up to one year after inclusion
  Clinical, neurophysiological and radiological evaluation of the lesions in question.
Time to disappearance of hemorrhages. | Up to three months after inclusion
Time to disappearance of paresis and/or paresthesias. | Up to one year after inclusion
Time to disappearance of pain. | Up to one year after inclusion
Time to disappearance of pulmonary infiltrates | Up to one month after inclusion
  Disappearance of inflammatory processes in the lung.
Time to disappearance of oxygen supplementation | Up to one month after inclusion
Incidence of severe infections | Up to one year after inclusion
  Incidence of severe bacterial, viral and fungal infections.
Incidence of graft versus host disease | Up to one year after inclusion
Actuarial survival | Up to 5 years after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Olle Ringdén, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Stockholm County, Sweden